CLINICAL TRIAL: NCT00858468
Title: Proof of Concept Study of the Safety and Immunogenicity of Influenza Virus Vaccine Fluzone® 2004-2005 Among Healthy Children 2 Months vs 6 Months of Age
Brief Title: Safety and Immunogenicity Testing of Influenza Vaccine in Healthy Children 2 Months and 6 Months of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC27
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2009-07-31 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Participants aged 6 to 12 Weeks at enrollment
  Interventions: Biological: Influenza virus vaccine (2004-2005 Formulation)
- Group 2 (Experimental): Participants aged 24 to 36 Weeks at enrollment
  Interventions: Biological: Influenza virus vaccine (2004-2005 Formulation)

INTERVENTIONS:
Biological: Influenza virus vaccine (2004-2005 Formulation) — 0.25 mL, Intramuscular
  Other Names: Fluzone® Preservative-free
  Arms: Group 1
Biological: Influenza virus vaccine (2004-2005 Formulation) — 0.25 mL, Intramuscular
  Other Names: Fluzone® Preservative-free
  Arms: Group 2

SUMMARY:
Primary Objective:

To describe the safety of the 2004-2005 pediatric formulation of the inactivated, split-virion influenza vaccine Fluzone®, given in the two-dose schedule (described in the package insert for vaccine-naïve young children) to the investigational and control groups.

Observational Objective:

To describe the percentage of protective Hemagglutination Inhibition (HAI) antibody titers (following a 2-dose Fluzone® immunization series) to each of the 3 vaccine antigens among the investigational and control groups.

DETAILED DESCRIPTION:
This is an observational and descriptive study that will provide preliminary comparative information about the safety and immunogenicity of Fluzone® vaccine among children aged 6 to 12 weeks (the investigational group, also referred to as the 2-month-old group) versus children aged 24 to 36 weeks (the control group, also referred to as the 6-month-old group). The study is not designed to achieve any preset statistical power, and no hypotheses will be tested.

ELIGIBILITY:
Inclusion Criteria :

* Aged 42 to 84 days (6 to 12 weeks) or 24 to 36 weeks on the day of inclusion.
* Born at full term of pregnancy (≥ 36 weeks) with a birth weight ≥ 2.5 kg.
* Considered to be in good health on the basis of reported medical history and history-directed physical examination.
* Available for the duration of the study.
* Parent/guardian willing and able to provide informed consent.
* Parent/guardian able to attend all scheduled visits and comply with all trial procedures.
* Willingness to permit venipuncture or heel stick for purposes of collecting a blood sample.

Exclusion Criteria :

* Reported allergy to egg proteins, chicken proteins or any other constituent of the vaccine.
* Previous history of influenza vaccination or documented history of influenza infection.
* Receipt of any vaccine in the 7 days prior to enrollment.
* An acute illness with fever (rectal temperature ≥ 38.0 °C [or ≥ 100.4 °F]) in the 72 hours preceding enrollment in the trial (defer enrollment).
* Known bleeding disorder.
* Participation in any other clinical trial within 30 days prior to enrollment, or planned participation in another clinical trial prior to termination of the subject's participation in this study.
* Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital or developmental disorder that could interfere with trial conduct or completion.
* Known HIV-positive or HBsAg-positive mother.
* Known HIV, hepatitis B (HBsAg), or hepatitis C infection.
* Blood or blood-derived products received in the past 2 months.
* Prior history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 2 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 394 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (8):
- United States (8):
  - Little Rock, Arkansas
  - Marietta, Georgia
  - Durham, North Carolina
  - Akron, Ohio
  - Dayton, Ohio
  - Pittsburgh, Pennsylvania
  - Norfolk, Virginia
  - Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 08 April to 05 August 2005 in 8 medical centers in the US
Pre-assignment Details: A total of 394 participants that met the inclusion and exclusion criteria were enrolled, 393 were vaccinated.
Groups:
- Age 6 to 12 Weeks: Participants enrolled at 6 to 12 weeks of age
- Age 24 to 36 Weeks: Participants enrolled at 24 to 36 weeks of age
Period: Overall Study
Arm/Group | Age 6 to 12 Weeks | Age 24 to 36 Weeks
Started | 201 (1 enrolled participant was not vaccinated and removed from analysis) | 192
Completed | 201 | 192
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 6 to 12 Weeks | Age 24 to 36 Weeks | Total
Number analyzed (Participants) | 201 | 192 | 393
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 201 | 192 | 393
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.4 (0.98) | 27.0 (1.31) | 18.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 99 | 197
  Male | 103 | 93 | 196
Region of Enrollment [Number; unit: participants]
  United States | 201 | 192 | 393

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local and Systemic Reactions After Vaccination With Fluzone® 2004-2005 Pediatric Formulation.
Description: Solicited local (injection site) reactions: Tenderness, erythema (redness), and swelling Solicited systemic reactions: Fever (Temperature), Vomiting, Crying abnormal, Drowsiness, Loss of Appetite, and Irritability.
Time Frame: Day 0 to Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intend-to-treat population
Measure: Number; unit: Percentage of participants
Arm/Group | Age 6 to 12 Weeks | Age 24 to 36 Weeks
Number analyzed (Participants) | 201 | 192
Percentage of participants
  Any Solicited Injection Site Reaction - Dose 1 | 54 | 47
  Any Tenderness | 50 | 44
  Grd 3 Tenderness-Inj. Limb movement reduced | 6 | 2
  Any Redness | 11 | 7
  Grade 3 Redness (≥ 5.0 cm) | 0 | 0
  Any Swelling | 8 | 5
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Injection Site Reaction - Dose 2 | 41 | 27
  Any Tenderness | 38 | 26
  Grd 3 Tenderness-Inj. Limb movement reduced | 1 | 0
  Any Redness | 10 | 5
  Grade 3 Redness (≥ 5.0 cm) | 1 | 0
  Any Swelling | 5 | 2
  Grade 3 Swelling (≥5.0 cm) | 0 | 0
  Any Solicited Injection Site Reaction - Any Doses | 61 | 52
  Any Tenderness | 57 | 50
  Grd 3 Tenderness-Inj. Limb movement reduced | 7 | 2
  Any Redness | 16 | 10
  Grade 3 Redness (≥ 5.0 cm) | 1 | 0
  Any Swelling | 12 | 6
  Grade 3 Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Systemic Reaction Dose 1 | 90 | 82
  Any Fever (Rectal Temp) | 8 | 18
  Grade 3 Fever (>39.5 ºC) | 0 | 0
  Any Vomiting | 22 | 16
  Grade 3 Vomiting (≥ 6 episodes per 24 hrs) | 1 | 0
  Any Abnormal Crying | 59 | 45
  Grade 3 Abnormal Crying | 3 | 3
  Any Drowsiness | 72 | 50
  Grade 3 Drowsiness (difficulty waking up) | 2 | 1
  Any Loss of Appetite | 43 | 35
  Grd 3 Loss of Appetite (refuses ≥ 3 meals) | 0 | 2
  Any Irritability | 77 | 67
  Grade 3 Irritability (inconsolable) | 5 | 3
  Any Solicited Systemic Reaction Dose 2 | 70 | 70
  Any Fever (Rectal Temp) | 4 | 14
  Grade 3 Fever (>39.5 ºC) | 0 | 2
  Any Vomiting | 14 | 8
  Grade 3 Vomiting (≥ 6 episodes per 24 hrs) | 1 | 0
  Any Abnormal Crying | 37 | 34
  Grade 3 Abnormal Crying | 4 | 1
  Any Drowsiness | 47 | 38
  Grade 3 Drowsiness (difficulty waking up) | 2 | 0
  Any Loss of Appetite | 28 | 27
  Grade 3 Loss of Appetite (refuses ≥ 3 meals) | 1 | 0
  Any Irritability | 55 | 53
  Grade 3 Irritability (inconsolable) | 3 | 1
  Any Solicited Systemic Reaction Any Dose | 92 | 89
  Any Fever (Rectal Temp) | 11 | 26
  Grade 3 Fever (>39.5 ºC) | 0 | 2
  Any Vomiting | 27 | 21
  Grade 3 Vomiting (≥ 6 episodes per 24 hrs) | 2 | 0
  Any Abnormal Crying | 66 | 55
  Grade 3 Abnormal Crying | 6 | 4
  Any Drowsiness | 78 | 58
  Grade 3 Drowsiness (difficulty waking up) | 4 | 1
  Any Loss of Appetite | 52 | 47
  Grade 3 Loss of Appetite (refuses ≥ 3 meals) | 1 | 2
  Any Irritability | 82 | 76
  Grade 3 Irritability (inconsolable) | 7 | 4

2. Other Pre Specified Outcome: Percentage of Participants With Serum Hemagglutination Inhibition Antibody Titer ≥ 40 Post-vaccination With Fluzone® (Seroprotection).
Description: Data presented for each of the three influenza vaccine virus antigens in the Fluzone® 2004-2005 pediatric formulation.
  Seroprotection was defined as the percentage of participants with a reciprocal hemagglutination inhibition titers ≥ 40
Time Frame: 21 days post-vaccination 2
Population: Seroprotection analysis was in all enrolled and vaccinated participants in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of participants
Arm/Group | Age 6 to 12 Weeks | Age 24 to 36 Weeks
Number analyzed (Participants) | 149 | 144
Percentage of participants
  A/NEW CALEDONIA/20/99 ≥ 40 Post-dose | 46 | 69
  A/WYOMING/03/2003 ≥ 40 Post-dose | 59 | 78
  B/JIANGSU/10/2003 ≥ 40 Post-dose | 5 | 22

3. Other Pre Specified Outcome: Percentage of Participants With a Pre-vaccination Serum Hemagglutination Inhibition Antibody Titer of ≤ 10 That Had a Titer of ≥ 40 Post-vaccination With Fluzone® (Seroconversion).
Description: Seroconversion was defined as the percentage of participants with a pre-titer < 1:10 who demonstrated a ≥ 4-fold increases in titer from pre- to post-vaccination.
Time Frame: 21 days post-vaccination 2
Population: Seroconversion analysis was in all enrolled and vaccinated participants in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of participants
Arm/Group | Age 6 to 12 Weeks | Age 24 to 36 Weeks
Number analyzed (Participants) | 149 | 144
Percentage of participants
  A/NEW CALEDONIA/20/99, Pre-Dose ≤ 10 | 70 | 96
  A/NEW CALEDONIA/20/99, Pre-Dose ≤10, Post-Dose ≥40 | 48 | 72
  A/WYOMING/03/2003, Pre-Dose ≤ 10 | 32 | 74
  A/WYOMING/03/2003, Pre-Dose ≤10, Post-Dose ≥40 | 60 | 86
  FLU B/JIANGSU/10/2003, Pre-Dose ≤ 10 | 84 | 97
  FLU B/JIANGSU/10/2003, Pre-Dose ≤10, Post-Dose ≥40 | 4 | 20

4. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Antibodies Pre- and Post-vaccination With Fluzone® Vaccine.
Description: Data presented for each of the three influenza vaccine virus antigens in the Fluzone® 2004-2005 pediatric formulation.
Time Frame: 21 days post-vaccination 2
Population: GMTs were assessed on the Per-Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Age 6 to 12 Weeks | Age 24 to 36 Weeks
Number analyzed (Participants) | 149 | 144
Titers
  A/NEW CALEDONIA/20/99 Pre-dose | 11.5 [9.4 to 14.1] | 5.7 [5.3 to 6.0]
  A/NEW CALEDONIA/20/99 Post-dose | 27.6 [23.1 to 33.1] | 47.0 [39.3 to 56.2]
  A/WYOMING/03/2003 Pre-dose | 40.8 [31.2 to 53.2] | 9.8 [8.1 to 11.9]
  A/WYOMING/03/2003 Post-dose | 46.3 [38.7 to 55.4] | 90.9 [72.2 to 114.4]
  B/JIANGSU/10/2003 Pre-dose | 7.0 [6.3 to 7.8] | 5.4 [5.1 to 5.7]
  B/JIANGSU/10/2003 Post-dose | 8.4 [7.5 to 9.3] | 15.3 [12.9 to 18.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months post-vaccination.
Arm/Group | Age 6 to 12 Weeks | Age 24 to 36 Weeks
Serious Adverse Events (participants affected / at risk) | 4/201 | 3/192
Other Adverse Events (participants affected / at risk) | 54/201 | 94/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 6 to 12 Weeks (N=201) | Age 24 to 36 Weeks (N=192)
Kawasaki's disease (Infections and infestations) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (3)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 6 to 12 Weeks (N=201) | Age 24 to 36 Weeks (N=192)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 12 (13)
Teething (Gastrointestinal disorders) | 0 (0) | 17 (22)
Injection site haemorrhage (General disorders) | 4 (5) | 10 (11)
Pyrexia (General disorders) | 5 (6) | 19 (20)
Nasopharyngitis (Infections and infestations) | 2 (2) | 11 (12)
Otitis media (Infections and infestations) | 3 (3) | 16 (18)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 19 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 16 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 15 (17)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications